CLINICAL TRIAL: NCT02588612
Title: A Pilot Open-Label Clinical Trial Evaluating the Safety and Efficacy of Autologous T Cells Expressing Enhanced TCRs Specific for NY-ESO-1 in Subjects With Stage IIIb or Stage IV Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Letetresgene Autoleucel Engineered T Cells in NY-ESO -1 Positive Advanced Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 208749; ADP-0011-004 (Other: Adaptimmune Therapeutics); 2016-002517-21 (EudraCT Number)
Record Dates: First submitted 2015-10-26; First posted 2015-10-28 (Estimated); Results first posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Neoplasms
Keywords: Letetresgene autoleucel; Adoptive TCR T-cell therapy; NY-ESO-1; T Cell Receptor; Non-Small Cell Lung Cancer; Leukapheresis
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- letetresgene autoleucel (GSK3377794) (Experimental): Eligible participants will be leukapheresed to manufacture engineered T-cells. Participants will then receive letetresgene autoleucel (GSK3377794), as a single intravenous (IV) infusion after completing lymphodepleting chemotherapy.
  Interventions: Drug: letetresgene autoleucel (GSK3377794); Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Drug: letetresgene autoleucel (GSK3377794) — letetresgene autoleucel (GSK3377794) as an IV infusion.
Drug: Cyclophosphamide — Cyclophosphamide will be used as a lymphodepleting chemotherapy.
Drug: Fludarabine — Fludarabine will be used as a lymphodepleting chemotherapy.

SUMMARY:
This trial will evaluate safety and efficacy of letetresgene autoleucel (GSK3377794) in participants with metastatic NSCLC.

DETAILED DESCRIPTION:
New York esophageal antigen-1 (NY-ESO-1) and L antigen family member (LAGE)-1a antigens are tumor-associated proteins that have been found in several tumor types. Clinical trials using adoptively transferred T-cells directed against NY-ESO-1/LAGE-1a have shown objective responses. Letetresgene autoleucel (GSK3377794) is the first generation of NY-ESO-1 specific T-cell receptor engineered TCR T-cells. This protocol investigates letetresgene autoleucel treatment in Human Leukocyte Antigen (HLA)*-A*02+ participants with NY-ESO1+ advanced metastatic non-small cell lung cancer as second line treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participant is >=18 years of age on the day of signing informed consent.
* Participant has a diagnosis of histologically or cytologically confirmed advanced non-small cell lung cancer (Stage IIIB or IV) or recurrent disease.
* Participants with known epidermal growth factor receptor (EGFR) mutations or Anaplastic lymphoma kinase receptor (ALK) or ROS1 gene rearrangements must have failed (disease progression [PD] or unacceptable toxicity) prior EGFR or ALK or ROS1 tyrosine kinase inhibitor, respectively (PD or unacceptable toxicity). There is no limit to lines of prior anti-cancer therapy.
* Participant has measurable disease according RECIST v1.1 criteria.
* Participant is HLA-A*02:01, HLA-A*02:05 and/or HLA-A*02:06 positive.
* Participant's tumor is positive for NYESO and/or LAGE-1a expression by a designated central laboratory.
* Participant has Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1.
* Participant has an anticipated life expectancy >3 months.
* Participant has left ventricular ejection fraction >=50 percent(%).
* Participant is fit for leukapheresis and has adequate venous access for the cell collection.
* Male or Female. Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Participant must have adequate organ function.

Exclusion Criteria:

* Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones, liver metastases or otherwise stable chronic liver disease per Investigator assessment).
* Washout periods for prior radiotherapy and chemotherapy and other systemic therapy must be followed.
* Experimental anti-cancer vaccine within 2 months prior to leukapheresis in the absence of response or in the opinion of the Investigator is responding to an experimental vaccine given within 6 months prior to leukapheresis.
* Any prior gene therapy using an integrating vector.
* Toxicity from previous anti-cancer therapy that has not recovered to less than or equal to (<=)Grade 1 prior to enrollment (with exceptions).
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cyclophosphamide, fludarabine, or other agents used in the study.
* Central nervous system (CNS) metastases.
* Active brain metastases or leptomeningeal metastases.
* History of chronic or recurrent (within the last year prior to enrollment) severe autoimmune or active immune-mediated disease requiring steroids or other immunosuppressive treatments.
* Other active malignancies besides NSCLC within 3 years prior to Screening not in complete remission.
* Unintended weight loss >10% in 6 months preceding study entry.
* Corrected QT interval (QTc) >450 milliseconds (msec) or QTc >480 msec for participants with Bundle Branch Block (BBB).
* Uncontrolled intercurrent illness.
* Participants who in the opinion of the Investigator will be unlikely to fully comply with protocol requirements.
* Active infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV) or human T-cell lymphotropic virus (HTLV).
* Participant is pregnant or breastfeeding.
* Major surgery within 4 weeks prior to lymphodepleting chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2020-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (3):
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label study evaluating the safety and tolerability of autologous T-Cells expressing enhanced T-cell receptors (TCRs) specific for New York esophageal squamous cell carcinoma (NY-ESO)-1 (letetresgene autoleucel, lete-cel, GSK3377794) in Human Leukocyte Antigen (HLA)-A*02:01, HLA-A*02:05 and/or HLA-A*02:06 participants with stage IIIb or stage IV non-small cell lung cancer (NSCLC).
Pre-assignment Details: Participants were screened for the specified HLA alleles and target antigen expression (NY-ESO-1), and evaluated for study eligibility. A total of 10 participants who met all the eligibility criteria were enrolled in this study which consisted of Intent-to-Treat (ITT) population. This study was conducted across 3 sites in the United States.
Groups:
- Lete-cel: Eligible participants were leukapheresed to manufacture lete-cel. Participants then underwent lymphodepleting chemotherapy with cyclophosphamide and fludarabine followed by a single intravenous (IV) infusion of lete-cel.
Period: Overall Study
Arm/Group | Lete-cel
Started | 10
Received T-cell Infusion | 5
Completed | 5
Not Completed | 5
Not completed — Physician Decision | 1
Not completed — Leukapheresis did not yield enough cells | 1
Not completed — Failed eligibility prior to chemotherapy | 2
Not completed — Death prior to T-cell infusion | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lete-cel
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Overall study | 57.7 (12.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  White | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Non-serious Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or is clinically significant or requires intervention to prevent one of the outcomes listed before. Number of participants with common (greater than or equal to [>=]5 percent[%]) non-serious AEs and SAEs are presented.
Time Frame: Up to 24 months
Population: ITT population consisted of all participants who were enrolled in the trial and met all eligibility criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Lete-cel
Number analyzed (Participants) | 10
Participants
  Non SAEs | 6
  SAEs | 4

2. Primary Outcome: Number of Participants With Hematology Results by Maximum Grade Increase Post-Baseline
Description: Blood samples were collected for the analysis of following hematology parameters: hemoglobin, lymphocytes, neutrophils, platelets and leukocytes. Laboratory parameters were graded according to National Cancer Institute-Common Toxicity Criteria for Adverse Events (NCI-CTCAE) version 4.03 where, Grade1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. Baseline is the most recent, non-missing value from a central laboratory within 7 days prior to the lymphodepleting chemotherapy. An increase in grade is defined as an increase in CTCAE grade relative to Baseline grade. Data for any grade increase at worst-case post-Baseline is presented
Time Frame: Up to 24 months
Population: Modified (m)ITT population consisted of all participants in the ITT population who received NYESO-1 T cell infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | Lete-cel
Number analyzed (Participants) | 5
Participants
  Hemoglobin increased | 0
  Hemoglobin (Anemia) | 3
  Lymphocytes increased | 1
  Lymphocytes decreased | 5
  Neutrophils | 5
  Platelets | 5
  Leukocytes (Leukocytosis) | 0
  Leukocytes (Leukopenia) | 5

3. Primary Outcome: Number of Participants With Any Grade Increase in Clinical Chemistry Parameters
Description: Blood samples were collected for analysis of clinical chemistry parameters: glucose (Gl), albumin, alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin (Bil), creatinine (Creat), potassium (Pot), magnesium (Mg), phosphate (Ph), sodium (Sod) and calcium. Laboratory parameters were graded according to NCI-CTCAE version 4.03 where, Grade1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. An increase in grade is defined as an increase in CTCAE grade relative to Baseline grade. Data for any grade increase at worst-case post-Baseline is presented.
Time Frame: Up to 24 months
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Lete-cel
Number analyzed (Participants) | 5
Participants
  Gl, Hyperglycemia | 2
  Gl, Hypoglycemia | 0
  Albumin | 2
  ALP | 2
  ALT | 3
  AST | 4
  Bil | 1
  Creat | 1
  Pot, Hyperkalemia | 2
  Pot, Hypokalemia | 1
  Mg, Hypermagnesemia | 0
  Mg, Hypomagnesemia | 2
  Ph | 4
  Sod, Hypernatremia | 0
  Sod, Hyponatremia | 1
  Calcium, Hypercalcemia | 1
  Calcium, Hypocalcemia | 3

4. Primary Outcome: Number of Participants With Worst Case Post-Baseline Abnormal Electrocardiogram (ECG) Findings
Description: 12-lead ECGs were recorded in semi-supine position after 5 minutes rest using an ECG machine that automatically calculated the heart rate and measured PR, RR, QRS and QT duration corrected for heart rate by Fridericia's formula (QTcF) intervals. Data for number of participants with abnormal not clinically significant (NCS) and clinically significant (CS) ECG findings for worst case post-Baseline have been presented. Clinically significant abnormal laboratory findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Up to 24 months
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Lete-cel
Number analyzed (Participants) | 5
Participants
  Abnormal, NCS | 2
  Abnormal, CS | 1

5. Primary Outcome: Change From Baseline in Oxygen Saturation
Description: Oxygen saturation measures the capacity of blood to transport oxygen to other parts of the body. Oxygen saturation was measured using a pulse oximeter. Baseline is the most recent, non-missing value within 7 days prior to initiating the lymphodepleting chemotherapy. Change from Baseline is the post-Baseline visit value minus Baseline value.
Time Frame: Baseline, Day 1 (pre-dose, 5, 15, and 30 minutes, 1, 1.5, 2, and 4 hours post dose), Days 2, 3, 4, 5, 8 and Week 2
Population: mITT Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in category titles).
Measure: Median (Full Range); unit: Percentage of oxygen
Arm/Group | Lete-cel
Number analyzed (Participants) | 5
Percentage of oxygen
  Day 1, pre dose, n=5 | 2.0 [-2 to 6]
  Day 1, 5 minutes post dose, n=4: number analyzed (Participants) | 4
  Day 1, 5 minutes post dose, n=4 | 2.5 [1 to 3]
  Day 1, 15 minutes post dose, n=4: number analyzed (Participants) | 4
  Day 1, 15 minutes post dose, n=4 | 2.0 [-3 to 5]
  Day 1, 30 minutes post dose, n=4: number analyzed (Participants) | 4
  Day 1, 30 minutes post dose, n=4 | 3.0 [-2 to 3]
  Day 1, 1 hour post dose, n=5 | 2.0 [-2 to 5]
  Day 1, 1.5 hours post dose, n=2: number analyzed (Participants) | 2
  Day 1, 1.5 hours post dose, n=2 | 1.5 [1 to 2]
  Day 1, 2 hours post dose, n=3: number analyzed (Participants) | 3
  Day 1, 2 hours post dose, n=3 | 3.0 [2 to 5]
  Day 1, 4 hours post dose, n=4: number analyzed (Participants) | 4
  Day 1, 4 hours post dose, n=4 | -1.0 [-3 to 3]
  Day 2, n=4: number analyzed (Participants) | 4
  Day 2, n=4 | 2.5 [1 to 4]
  Day 3, n=5 | 1.0 [-1 to 4]
  Day 4 , n=5 | 1.0 [-3 to 4]
  Day 5, n=5 | -2.0 [-3 to 4]
  Day 8, n=4: number analyzed (Participants) | 4
  Day 8, n=4 | 0.0 [-1 to 1]
  Week 2, n=4: number analyzed (Participants) | 4
  Week 2, n=4 | 1.5 [1 to 3]

6. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants with a confirmed Partial response (PR) or Complete response (CR) as the Best overall response (BOR), as assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1. Confidence Interval (CI) was calculated using the exact method. Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the Baseline sum diameters. Complete response is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 millimeters.
Time Frame: Up to 24 Months
Population: mITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lete-cel
Number analyzed (Participants) | 5
Percentage of participants | 20 [0.5 to 71.6]

7. Secondary Outcome: Time to Response
Description: Time to response is defined as the interval of time (in months) between the date of T-cell infusion and the first documented evidence of response (PR or CR) in the subset of participants with a confirmed PR or CR as the BOR as assessed by the investigator per RECIST v1.1.
Time Frame: Up to 24 months
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Number; unit: Months
Arm/Group | Lete-cel
Number analyzed (Participants) | 1
Months | 12.09

8. Secondary Outcome: Duration of Response
Description: Duration of response (DoR), defined as the interval of time in months from first documented evidence of PR or better to the time when disease progression is documented as assessed by RECIST v1.1 or death due to any cause among participants with a confirmed PR or CR as the BOR.
Time Frame: Up to 24 months
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Number; unit: Months
Arm/Group | Lete-cel
Number analyzed (Participants) | 1
Months | 6.18

9. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of participants with a stable disease (SD) or better as the BOR (Confirmed PR, confirmed CR, or SD >=12 weeks), as assessed by the investigator per RECIST v1.1. CI was calculated using the exact method.
Time Frame: Up to 24 months
Population: mITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lete-cel
Number analyzed (Participants) | 5
Percentage of participants | 20 [0.5 to 71.6]

10. Secondary Outcome: Progression-Free Survival (PFS) by Investigator Assessment
Description: Progression-free survival (PFS) is defined as the interval of time (in months) between the date of T-cell infusion and the earlier of the date of disease progression as assessed by the investigator and the date of death due to any cause. Progressive Disease (PD) is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. PFS based on responses assessed by investigator per RECIST v1.1 is presented. Median and inter-quartile range (first quartile and third quartile) are presented.
Time Frame: Up to 24 months
Population: mITT Population
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Lete-cel
Number analyzed (Participants) | 5
Months | 1.81 [0.99 to 5.29]

ADVERSE EVENTS:
Time Frame: All-cause mortality, SAEs and common (>=5%) non-serious AEs were collected from the enrollment to 24 months
Description: All-cause mortality, SAEs and common non-serious AEs were reported for the ITT Population which comprised of all participants enrolled in the study.
Arm/Group | Lete-cel
All-Cause Mortality (participants affected / at risk) | 4/10
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lete-cel (N=10)
Cytokine release syndrome (Immune system disorders) | 2
Pneumonia (Infections and infestations) | 2
Anaemia (Blood and lymphatic system disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lete-cel (N=10)
Lymphocyte count decreased (Investigations) | 5
White blood cell count decreased (Investigations) | 5
Neutrophil count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 4
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Anaemia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 2
Leukocytosis (Blood and lymphatic system disorders) | 1
Lymph node pain (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 3
Oedema peripheral (General disorders) | 2
Asthenia (General disorders) | 1
Chills (General disorders) | 1
Pyrexia (General disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 3
Lethargy (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Paralysis (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Supraventricular tachycardia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Bronchitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Strongyloidiasis (Infections and infestations) | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Confusional state (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 2
Urinary retention (Renal and urinary disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/12/NCT02588612/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-02): https://cdn.clinicaltrials.gov/large-docs/12/NCT02588612/SAP_001.pdf